CLINICAL TRIAL: NCT00001132
Title: A Pilot Study of Early Treatment Intensification of Antiretroviral Therapy
Brief Title: Effectiveness of the Early Addition of Abacavir to an Anti-HIV Drug Combination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG A5064; AACTG A5064
Record Dates: First submitted 2000-01-17; First posted 2001-08-31 (Estimated); Last update posted 2008-09-09 (Estimated); Status verified 2003-06

CONDITIONS: HIV Infections
Keywords: Placebos; HIV-1; Drug Therapy, Combination; RNA, Viral; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; abacavir
MeSH Terms: conditions — HIV Infections | interventions — abacavir

INTERVENTIONS:
Drug: Abacavir sulfate

SUMMARY:
The purpose of this study is to see if adding 1 drug to an anti-HIV drug combination early in treatment against HIV can lower the viral load (amount of HIV in the blood) to a level so low that it cannot be measured (undetectable). The drug that will be added to a treatment is abacavir (ABC).

Many patients who take 3 anti-HIV drugs together are able to achieve very low viral loads, for example, viral loads below 50 copies/ml. However, some patients taking only 3 drugs are not able to achieve a viral load this low. Doctors hope that, by adding the drug ABC to a current treatment, a viral load below 50 copies/ml can be achieved. Doctors would like to find out if it is effective to start patients on 3 drugs and then add another drug (treatment intensification) if the treatment is not working as well as hoped.

DETAILED DESCRIPTION:
Combination antiretroviral therapy can offer patients potent suppression of HIV replication and improved immunologic functioning. However, despite aggressive antiretroviral regimens currently in use, only about 50 to 60 percent of patients attain plasma viral loads below 50 copies/ml after 24 weeks. Initiating treatment with a 4-drug regimen may increase this percentage, but this may also contribute to patient non-adherence, drug-related toxicities, potential cross-resistance to drugs used in future regimens, and high financial costs. Another strategy is early intensification (adding a single drug to an existing regimen) in patients who are at risk for attaining incomplete viral suppression after 24 weeks of therapy. ABC may produce a significant antiviral effect when used as an intensification agent in patients on a stable antiretroviral regimen. The results of this study will offer insight into the potential benefits of early treatment intensification.

Patients entering this study will have initiated potent antiretroviral therapy. Between 60 and 90 days [AS PER AMENDMENT 1/9/01: 60 and 104 days] after beginning their background regimen, patients are randomized to add either ABC (Arm A) or a matching placebo (Arm B) for 12 weeks. Patients completing 12 weeks of treatment continue on study for an additional 24 weeks to Week 36. Patients discontinue treatment if virologic failure occurs at any time. Patients still return to the clinic for HIV-1 RNA measurements at Weeks 12 and 36, depending on when discontinuation occurred. Patients who discontinue treatment at or after Week 12 due to virologic failure are offered open-label ABC for the remainder of the study (through Week 36). Blood samples are collected at Weeks 4, 8, 12, 20, 28, and 36. Plasma samples for population sequencing of HIV-1 PR and RT genes are collected on all patients at study entry and at the time of virologic failure. Baseline genotype (presence or absence of PR and RT resistance mutations and number of resistance mutations) is correlated to treatment outcome. Samples from the time of failure are analyzed for the accumulation of additional resistance mutations. [AS PER AMENDMENT 5/5/00: Patients and their primary care physicians will be unblinded to the patient's treatment after the study is completed at Week 36 or if virologic failure occurs at or after Week 12 [AS PER AMENDMENT 1/9/01: or if ABC hypersensitivity is suspected].]

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have been taking anti-HIV therapy that includes at least 3 anti-HIV drugs and is an acceptable anti-HIV drug combination for 60 to 104 days before study treatment. Patients must not have changed any of the drugs in the 28 days before study entry. (This study has been changed by extending the number of days that anti-HIV therapy has been received.)
* Have a viral load greater than 500 but less than or equal to 10,000 copies/ml and have had a significant decrease in viral load between 49 and 84 days after starting this anti-HIV therapy. (This study has been changed by extending the length of time of viral load decrease.)
* Are at least 13 years old (consent of parent or guardian required if under 18).
* Agree to practice abstinence or use barrier method of birth control (such as condoms) during the study and for 3 months after.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have ever taken ABC.
* Have received anti-HIV therapy for more than 104 days in the past. (This study has been changed by extending the number of days that anti-HIV therapy has been received.)
* Have a fever for 7 days in the 30 days before study entry.
* Have cancer, including Kaposi's sarcoma, that requires chemotherapy.
* Have an active infection that requires treatment in the 21 days before study entry.
* Have any opportunistic (AIDS-related) infection or disease that requires a change in medication in the 14 days before study entry.
* Have any medical condition or history of an illness that the doctor feels would place them at risk or make them unable to complete the study.
* Are taking drugs that affect the immune system or any experimental anti-HIV drugs, except for their current drug combination.
* Are taking St. John's wort. (This study has been changed. Previously, patients taking St. John's wort were eligible.)
* Have received a vaccine in the 21 days before study entry.
* Are pregnant or breast-feeding.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Start 1999-11; Study Completion 2001-04

CONTACTS AND LOCATIONS:
Overall Officials: John Bartlett, Study Chair; Pablo Tebas, Study Chair
Locations (30):
- United States (29):
  - UCLA CARE Ctr, Los Angeles, California
  - Willow Clinic, Menlo Park, California
  - Santa Clara Valley Med Ctr / AIDS Community Rsch Consortium, San Jose, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Univ of Miami School of Medicine, Miami, Florida
  - Emory Univ, Atlanta, Georgia
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - State of MD Div of Corrections / Johns Hopkins Univ Hosp, Baltimore, Maryland
  - Johns Hopkins Hosp, Baltimore, Maryland
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Aaron Diamond AIDS Rsch Ctr / Rockefeller Univ, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Philadelphia Veterans Administration Med Ctr, Philadelphia, Pennsylvania
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Univ of Texas, Southwestern Med Ctr of Dallas, Dallas, Texas
  - Univ of Washington, Seattle, Washington
- Univ of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Background] Bartlett JA, Tebas P, Bassett R, Huang W, Kuritzkes D, Reisler R, Loyack N, Robison K; ACTG A5064 Team. Early intensification with abacavir in subjects at high risk for incomplete viral suppression. Antivir Ther. 2003 Aug;8(4):361-3. No abstract available. PMID 14518706